CLINICAL TRIAL: NCT04314518
Title: The Correlation Between Immunological Reaction of the Seminal Fluid in the Mother's Blood and Pregnancy Complications
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-19-6226-NH-CTIL
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2021-09

CONDITIONS: Preeclampsia; Pregnancy Complications; Insemination; Complication; Immune Tolerance; Paternal Exposure
Keywords: Preeclampsia; Artificial insemination; Seminal fluid; Maternal immune tolerance; Trophoblast; Vasculogenesis; Placentation; NK cells; T cells; Skin prick test
MeSH Terms: conditions — Pre-Eclampsia; Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — After enrollment, Seminal fluid sample will be extracted from the sperm sample of the donor at the sperm bank of Sheba medical center.
  After enrollment and in close proximity to the artificial insemination each woman will donate blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
It is known that if there isn't an efficient exposure to the paternal antigens before conception, there is an increased risk for the pre-eclampsia (PE) cascade and other pregnancy complications to take place.

It is possible that maternal immune system that doesn't develop tolerance to the paternal antigens that the seminal fluid carries, doesn't developed an adequate immune tolerance to the trophoblast cells and due to that, they are being under greater attack during placentation. Thus, the cells don't go through a normal differentiation, don't perform normal pseudo-vasculogenesis and the PE cascade is more likely to be carried out.

Both the maternal immune system and the paternal alloantigens have a role in the development of PE. Although the specific etiology remains unclear and can be only hypothesized.

In this study the investigators aim is to try and prove that there is a difference in the immunological reactions to semen prior to conception and that these changes are related to PE and/or other obstetric complications.

Hence the investigators aim to study the immune response to semen of women that will be exposed to the culprit semen for the first time compare to women that have been exposed to a culprit semen more than once previously (namely more than 1 insemination prior to the time of evaluation). After that, in a prospective cohort study the investigators would follow those women through their pregnancies and check for different pregnancy outcomes.

In this manner, the investigators are hoping to create a screening tool that will help to predict pregnancy and fetal complications before conception related to maternal immune responses of paternal antigens.

DETAILED DESCRIPTION:
The pathophysiology of preeclampsia (PE) likely involves both maternal and fetal/placental factors. It has been established that poor placentation followed by oxidative stress/inflammation and abnormalities in the development of placental vasculature early during pregnancy may result in relative placental ischemia, which then leads to a release of antiangiogenic factors into the maternal circulation. Thus, it changes the maternal systemic endothelial function and cause hypertension and other manifestations of the disease.

Defects in spiral artery remodeling and trophoblast invasion, two related but separate processes, are characteristic of hypertensive disorders of pregnancy and fetal growth restriction. Still, the exact etiology of PE remains elusive.

In normal pregnancies, the cytotrophoblast cells of the developing placenta migrate through the decidua and part of the myometrium to invade both the endothelium and highly muscular tunica media of the maternal spiral arteries. In addition to that, they alter their adhesion molecule expression, a process referred to as pseudo-vasculogenesis.

By comparison, in PE, cytotrophoblasts fail to penetrate the myometrial segment and fail to go through pseudo-vasculogenesis.

Consequently, the spiral arteries fail to develop into large, tortuous vascular channels, resulting in placental hypoperfusion and ischemia. This defect in deep placentation has been associated with development of multiple adverse pregnancy outcomes like PE, fetal death, abruptio placentae, IUGR, Preterm labor etc.

One of the possible mechanisms responsible for defective trophoblast invasion of the spiral arteries is defective differentiation of trophoblasts. The focus on immunologic factors as a possible contributor to abnormal placental development was based, in part, upon the observation that prior exposure to paternal antigens is inversely correlated with the risk of preeclampsia. For instance, nulliparous women, women who change partners between pregnancies, have long interpregnancy intervals, use barrier contraception and conceive via intracytoplasmic sperm injection, all of which have less exposure to paternal antigens and a higher risk of developing PE. Moreover, there are also paternal contributions to PE such as a new partner, limited sperm exposure and the concept of a "dangerous father" (a father aged>45, obese and with a familial history of early-onset cardiovascular disease or hypertension). Last but not least, one of the most significant finding in this field is that donor sperm pregnancies (artificial insemination) which hold no pre-exposure to paternal antigens are much more likely to lead to PE.

In contrast, oral sex (with the father's baby) was found to protect against PE, a finding that from an immunological point of view due may be explained by the relatively greater exposure of sperm antigen to the mother immune system via the buccal mucosa.

Taking it all together the investigators assume that these putative risk factors cannot be entirely attributed to the maternal nor the paternal side, but to the encounter between those two. If there isn't an efficient exposure to the paternal antigens before conception, there is an increased risk for the PE cascade and other pregnancy complications to take place. This hypothesis can help in explaining the gap in the process that the investigators already described. It is possible that maternal immune system that doesn't develop tolerance to the paternal antigens that the seminal fluid carries, doesn't developed an adequate immune tolerance to the trophoblast cells and due to that, they are being under greater attack during placentation. Thus, they don't go through a normal differentiation, don't perform normal pseudo-vasculogenesis and the PE cascade is more likely to be carried out.

There are several immunological mechanisms that support this assumption:

* The interaction between NK cells and extra-villous trophoblast cells: In PE, conflict between maternal and paternal genes is believed to induce abnormal placental implantation through increased NK cell activity.
* HLA-G: A gene with few alleles, that can be found both in the placental interface and in the paternal seminal fluid, has a significant role in inhibiting maternal immune responses against foreign (paternal) antigens.
* Regulatory T cells (Treg): Much of present thinking seems to involve a critical role for Treg in maintaining immunological tolerance during pregnancy. It has been suggested that during evolution, a mechanism of extra-thymic differentiation of Treg emerged in the placental to enforce maternal-fetal tolerance.

Men has a clear evolutionary interest in ensuring that the immune system of his female partner accepts the semi-allogenic fetus. Due to that, he tries to "prime" the woman's immune system pre-conception.

In conclusion, it is well established that both the maternal immune system and the paternal alloantigens have a role in the development of PE. Although the specific etiology remains unclear and can be only hypothesized. Therapies should aim not to suppress the maternal immune tolerance system but rather to enhance tolerance.

In this study the investigators aim is to try and prove that there is a difference in the immunological reactions to semen prior to conception and that these changes are related to PE and/or other obstetric complications.

Hence the investigators aim to study the immune response to semen of women that will be exposed to the culprit semen for the first time compare to women that have been exposed to a culprit semen more than once previously (namely more than 1 insemination prior to the time of evaluation). After that, in a prospective cohort study the investigators would follow those women through their pregnancies and check for different pregnancy outcomes.

In this manner, the investigators are hoping to create a screening tool that will help to predict pregnancy and fetal complications before conception related to maternal immune responses of paternal antigens. If the investigators hypothesize turn out to be true, it can cause sperm banks all over the world to change their matching protocols and to test seminal fluid in the maternal blood sample before putting her through artificial insemination with a poor prognosis.

For the best of the investigator's knowledge evaluation of immunological reaction to paternal seminal fluid in the mother's blood prior conception has never been tried before.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45
* 50 women for each group.
* Primigravid or first insemination from a new partner/sperm donor (group I)
* Women exposed to sperm (from the same donor/partner ≥ 2 times) (Group II)
* Singleton gestation
* Obtained verbal/written consent to participate in study

Exclusion Criteria:

* o Multiple gestation

  * Multifetal gestation
  * Chronic hypertension
  * Chronic renal disease
  * Autoimmune disease (antiphospholipid syndrome, systemic lupus erythematosus)
  * Vascular disease
  * Pregestational diabetes mellitus

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Following immunological evaluation (as specified in sec. 3) we will prospectively follow the patients and record pregnancy outcomes. Women (from each group) will be divided into 2 sub-groups:
  1. PE pregnancies and other pregnancy complications
  2. Normal pregnancies In the end, we will compare between the groups and the immunology reactions at the beginning of the follow-up and see if there is a difference that is statistically significant based on the immunological results.
     * Women that are going through artificial insemination attend in routine follow ups in Sheba medical center that will allow continuation of follow up after the course of pregnancy.
     * Woman recruited to participate in the study will be marked as such by a "pop up" message appearing on their computerized medical file.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Pregnancy complications | 2 years (Anticipated)
  Pregnancy complications including PE, placental abruption, IUGR

SECONDARY OUTCOMES:
Other pregnancy complications (Clinical or sonographic) | 2 years (Anticipated)
  Sonographic indices of placental insufficiency, abortion, Intra uterine fetal death, Oligohidramnion, fetal anomalies, preterm delivery, preterm premature rupture of membranes, mode of delivery and conception success rates.

CONTACTS AND LOCATIONS:
Overall Officials: Natav Hendin, Medical student, Principal Investigator — Sheba Medical Center
Locations (2):
- Israel (2):
  - Sheba medical center, Ramat Gan
  - Tel Hashomer Hospital, Ramat Gan